CLINICAL TRIAL: NCT06517147
Title: Efficacy of Post Exercise Heat Stress Cooling Via Cyrogenx Body Cooling Device
Brief Title: Cooling Via Cryogenx Body Cooling Device
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brunel University (Other)
Responsible Party: Principal Investigator, Dr Oliver Gibson, Principal Investigator, Brunel University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 31870-A-Mar/2024- 50405-1
Record Dates: First submitted 2024-07-12; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Body Temperature Changes
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rate of change in core temperature during CRYOGENX cooling (Experimental): Participants will visit the laboratory on three occasions during this randomized, counter-balanced crossover study. The first visit will enable preliminary data collection and familiarisation to take place. The second and third visits will be experimental sessions (CRYOGENX cooling vs regular cooling), with the order of these randomised. The rate of change in core temperature during cooling observed in the two trials will be compared by paired sample t-tests.
  Interventions: Device: Cryogenx cooling
- Rate of change in core temperature during regular cooling (Experimental): Participants will visit the laboratory on three occasions during this randomized, counter-balanced crossover study. The first visit will enable preliminary data collection and familiarisation to take place. The second and third visits will be experimental sessions (CRYOGENX cooling vs regular cooling), with the order of these randomised. The rate of change in core temperature during cooling observed in the two trials will be compared by paired sample t-tests.
  Interventions: Device: Regular cooling

INTERVENTIONS:
Device: Cryogenx cooling — During the cooling phase of both trials established field based cooling approaches e.g., temperate temperature water spraying (30°C, 5 mL.min-1), and air circulation (electric fan 2 m distance, 1.7 m.s-1 will be implemented. During the CRYOGENX cooling trial, the product will be affixed to the participant's torso in accordance with manufacturer's instructions and they will receive cooling via this intervention in addition to water spraying and air circulation. During the control visit, no intervention will be applied however water spraying and air circulation will be received.
  Arms: Rate of change in core temperature during CRYOGENX cooling
Device: Regular cooling — During the cooling phase of both trials established field based cooling approaches e.g., temperate temperature water spraying (30°C, 5 mL.min-1), and air circulation (electric fan 2 m distance, 1.7 m.s-1 will be implemented. During the CRYOGENX cooling trial, the product will be affixed to the participant's torso in accordance with manufacturer's instructions and they will receive cooling via this intervention in addition to water spraying and air circulation. During the control visit, no intervention will be applied however water spraying and air circulation will be received.
  Arms: Rate of change in core temperature during regular cooling

SUMMARY:
The aim of this project is to test the rate of cooling following exercise in the heat utilising the CRYOGENX Cryosuit device i) against passive cooling, and ii) to quantify the rate of cooling and compare this rate with established cooling intervention thresholds i.e. -0.11 to 0.15°C.min-1. As this project is to determine the efficacy of the intervention in populations equivalent to sporting and military personnel, these aims will be tested in young (18-40 year old) healthy male and female participants whom participate in regular physical activity. As a commercially funded project, the experimental design implemented will closely replicate that of the independent investigation into the efficacy of the CAERvest® device.

ELIGIBILITY:
The inclusion criteria are:

Aged 18 - 40 years Free from known injury, illness and disease and regular use of medications other than oral contraceptives Undertake exercise training >3 times per week for ~30 minutes per session

The exclusion criteria are:

Pregnant Previous history of neuromuscular fatigue Previous history of heat intolerance

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Core (rectal) temperature | 12 months
  The rate of change of core temperature during cooling will be calculated from realtime data

IPD SHARING:
Plan to Share IPD: Undecided